CLINICAL TRIAL: NCT01649700
Title: Treatment of Sequelae Caused by Severe Brain Injury With Autologous Adipose-derived Mesenchymal Stem Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Oscar Kuang-Sheng Lee, Director of Stem Cell Research Centre, National Yang Ming Chiao Tung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB-VGH-201101
Record Dates: First submitted 2012-04-09; First posted 2012-07-25 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: The Sequelae Caused by Severe Brain Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mesenchymal stem cells treatment (Experimental): All subjects will receive autologous adipose-derived mesenchymal stem cells
  Interventions: Biological: autologous adipose-derived mesenchymal stem cells

INTERVENTIONS:
Biological: autologous adipose-derived mesenchymal stem cells — Patients will receive five infusions, one month apart, each comprising 5-7x10^7 cells of autologous adipose-derived mesenchymal stem cells.

SUMMARY:
The study is to investigate the efficacy and safety of autologous transplantation of adipose-derived mesenchymal stem cells in patients with the sequelae caused by severe brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed diagnosis of a brain AVM (arteriovenous malformation).
* Stroke-like symptoms, including paralysis, caused by brain AVM hemorrhage.
* Subject's modified Rankin scale (mRS) grades IV~V.
* Ages between 20~40 years.
* Estimated life expectancy must be greater than 2 months.
* Signed informed consent from the subject.

Exclusion Criteria:

* Pregnancy test positive.
* Subject infected with hepatitis C, HIV or syphilis.
* Subject not suitable for liposuction surgery.
* Subject not eligible for PET or MRI.
* Subject enrolled in any other cell therapy studies within the past 30 days.
* Subject deemed to be not suitable for the study by the investigator.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety evaluation | 16 months
  Safety evaluate through vital signs, the results of clinical lab tests and adverse events (AEs).

SECONDARY OUTCOMES:
Positron emission tomography | 13 months
  18F-FDG used for the assessment of glucose metabolism in the brain
Magnetic Resonance Imaging | 16 months
  changes in the volume of brain lesions
Electroencephalogram | 16 months
  improvement of continuous slow-waves and irritative features
Neuropsychological assessment | 16 months
Electrodiagnostic Testing | 16 months
  improvement of subjects' sensory neurologic pathways
Assessment of language and swallowing functions | 16 months
  changes in levels of severity: normal/slight/mild/moderate/severe
Measure of the severity of disability | 16 months
Assessment of spasticity and strength | 16 months
Assessment of brain motor control | 16 months
  measurement of the electrical activities in the muscles during specific testing procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan